CLINICAL TRIAL: NCT00549575
Title: L-Arginine Treatment for Severe Vascular Fetal Intrauterine Growth Restriction: a Randomized Double Bind Controlled Trial
Brief Title: L-Arginine Treatment for Severe Vascular Fetal Intrauterine Growth Restriction: a Randomized Double Bind Controlled Trial (L Arginine in IUGR)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated
Sponsor: Nantes University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 99/4-A
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2007-10-26 (Estimated); Status verified 2007-10

CONDITIONS: Intra Uterine Growth Retardation
Keywords: Severe Intra uterine growth retardation below the third centile with abnormal uterine doppler; Severe growth retardation with pathologic uterine Doppler; L-Arginine; Nitric Oxide Donor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): Patients received 14 g/day of L-arginine (90 mL syrup, Veyron France Laboratories). Doppler ultrasound examination of the uterine, umbilical and cerebral circulation, and of ductus venous was performed prior to inclusion, after 7 days of treatment, and the day before delivery. Ultrasound examination was performed upon randomization, and weekly until birth. Venous blood and urine samples were collected before initiation and after 7 days of treatment, and both maternal and umbilical venous samples were obtained at delivery for nitrate and nitrite (NO2-/ NO3-) determination.
  Interventions: Drug: L ARG
- B (Placebo Comparator): After double blind randomization, patients received a placebo. Doppler ultrasound examination of the uterine, umbilical and cerebral circulation, and of ductus venous was performed prior to inclusion, after 7 days of treatment, and the day before delivery. Ultrasound examination was performed upon randomization, and weekly until birth. Venous blood and urine samples were collected before initiation and after 7 days of treatment, and both maternal and umbilical venous samples were obtained at delivery for nitrate and nitrite (NO2-/ NO3-) determination.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L ARG — Patients received 14 g/day of L-arginine (90 mL syrup, Veyron France Laboratories).
  Arms: A
Drug: Placebo — After double blind randomization, patients received a placebo.
  Arms: B

SUMMARY:
Although there is a strong rationale to supplement gravid patients suffering intrauterine growth restriction (IUGR) or preeclampsia with Arginine or other nitric oxide donors, evidence in the literature has been inconclusive. The current study was designed to determine whether oral treatment with L-Arginine, a nitric oxide (NO) donor, would enhance birth weight and/or decrease neonatal morbidity in pregnancies with severe vascular intrauterine growth restriction (IUGR).

DETAILED DESCRIPTION:
Patients and Methods: 44 patients with a singleton pregnancy who had been referred for IUGR detected by ultrasonic examination were included. Vascular IUGR was defined by fetal abdominal circumference less than or equal to the third percentile, associated with abnormal uterine Doppler. After double blind randomization, patients received either 14 g/day of L-arginine (90 mL syrup, Veyron France Laboratories), or a placebo. Doppler ultrasound examination of the uterine, umbilical and cerebral circulation, and of ductus venosus was performed prior to inclusion, after 7 days of treatment, and the day before delivery. Ultrasound examination was performed upon randomization, and weekly until birth. Venous blood and urine samples were collected before initiation and after 7 days of treatment, and both maternal and umbilical venous samples were obtained at delivery for nitrate and nitrite (NO2-/ NO3-) determination.

ELIGIBILITY:
Inclusion Criteria:

* Multicenter randomized trial.
* Patients with a singleton pregnancy with IUGR defined by fetal abdominal circumference less than or equal to the third percentile for gestational age, and abnormal uterine Doppler. Uterine Doppler was considered pathologic if Pourcelot's resistance index (S-D/S) was equal to or higher than 0.7, and/or if an obvious notch was present. If the placenta was not median, the side of the pathologic Doppler had to be on the same side as the placenta

Exclusion Criteria:

* Acute fetal distress
* Non vascular and non severe IUGR (normal uterine doppler scans and/or abdominal circumference > 3rd percentile)
* Maternal immune disorder
* IUGR from an infectious etiology
* IUGR associated with fetal malformation, multifetal pregnancy, and preeclampsia upon inclusion

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2000-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The principal outcome is birth weight at delivery and neonatal morbidity (Crib Score) | 6 weeks

SECONDARY OUTCOMES:
Secondary outcomes are Maternal and fetal hemodynamic with blood pressure and dopplers upon inclusion, after 7 days of treatment and at delivery | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Winer, Doctor, Principal Investigator — Nantes University Hospital; Dominique Darmaun, Professor, Study Chair — Nantes University Hospital; Philippe Gilard, Doctor, Study Chair — University Hospital, Angers; F Goffinet, Professor, Study Chair — Paris-Port-Royal
Locations (1):
- Chu-Nantes, Nantes, France

REFERENCES:
- [Derived] Winer N, Branger B, Azria E, Tsatsaris V, Philippe HJ, Roze JC, Descamps P, Boog G, Cynober L, Darmaun D. L-Arginine treatment for severe vascular fetal intrauterine growth restriction: a randomized double-bind controlled trial. Clin Nutr. 2009 Jun;28(3):243-8. doi: 10.1016/j.clnu.2009.03.007. Epub 2009 Apr 8. PMID 19359073